CLINICAL TRIAL: NCT04438798
Title: A Prospective Randomized Study of High Flow Nasal Cannula to Prevent Deoxygenation During Induction of General Anesthesia in Cesarean Section
Brief Title: High Flow Nasal Cannula to Prevent Deoxygenation During Induction of General Anesthesia in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0304665
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hypoxic Brain Injury; Maternal Death
MeSH Terms: conditions — Hypoxia, Brain; Maternal Death | interventions — Masks; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face mask group (Placebo Comparator): Pregnant females will be preoxygenated with 100% oxygen using a tight-fitting face mask at a rate of 6 L/min for 3 min with end-tidal gas monitoring.
  Interventions: Other: F Group
- THRIVE group (Active Comparator): High-flow humidified oxygen warmed to 37°C will be delivered through nasal cannula at the rate of 30 L/ min for 30 seconds then 50 liters per minute for a further 150 seconds.
  Interventions: Other: H Group

INTERVENTIONS:
Other: F Group — In Group F, pregnant females will be preoxygenated with 100% oxygen using a tight-fitting face mask at a rate of 6 L/min for 3 min with end-tidal gas monitoring.
  Other Names: face mask
  Arms: face mask group
Other: H Group — In Group H, high-flow humidified oxygen warmed to 37°C will be delivered through nasal cannula at the rate of 30 L/ min for 30 seconds then 50 liters per minute for a further 150 seconds.
  Other Names: THRIVE
  Arms: THRIVE group

SUMMARY:
Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) using high flow oxygen therapy for preoxygenation and oxygen supplementation during apnoea has shown promising results

DETAILED DESCRIPTION:
Eeffective preoxygenation followed by apnoeic oxygenation enables anaesthesiologists to safely prolong the apnoea time which is the time (seconds) of apnea following preoxygenation and muscle relaxation before to peripheral oxygen saturations (SpO2) decreases by 2%.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females
* Of American Society of Anesthesiologists (ASA) physical Status I and II
* For elective cesarean section under general anesthesia

Exclusion Criteria:

* with room air saturation of <98%
* anticipated difficult airway
* anticipated obstetric risk factor or precious baby
* chronic obstructive pulmonary disease
* thyrotoxicosis
* pheochromocytoma
* hyperkalaemia
* significant cardiac illness

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
measure the time of safe apnea | 10 minutes after induction
  The apnea time will start from the onset of cessation of breathing as evidenced by a flat line in the capnogram with the absence of chest movements

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Egypt

REFERENCES:
- [Background] Mir F, Patel A, Iqbal R, Cecconi M, Nouraei SA. A randomised controlled trial comparing transnasal humidified rapid insufflation ventilatory exchange (THRIVE) pre-oxygenation with facemask pre-oxygenation in patients undergoing rapid sequence induction of anaesthesia. Anaesthesia. 2017 Apr;72(4):439-443. doi: 10.1111/anae.13799. Epub 2016 Dec 30. PMID 28035669